CLINICAL TRIAL: NCT00443963
Title: Effects of Esomeprazole Magnesium on Gastric Free Radical Production and Total Antioxidant Capacity in Dyspeptic Patients Receiving Non-steroidal Anti-inflammatory Drugs
Brief Title: Total Antioxidant Effects of Esomeprazole in Dyspeptic Patients Receiving Non-steroidal Anti-inflammatory Drugs
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was not approved by the Human Studies Subcommittee.
Sponsor: Medstar Health Research Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Timothy Koch, Principal Investigator, Medstar Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRUSESOM0391
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Dyspepsia
Keywords: Dyspepsia in patients taking NSAIDs
MeSH Terms: conditions — Dyspepsia | interventions — Esomeprazole; Ranitidine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- PPI (Experimental): PPI Medication
  Interventions: Drug: Esomeprazole Magnesium
- H2RA (Experimental): H2RA Medication
  Interventions: Drug: Esomeprazole Magnesium

INTERVENTIONS:
Drug: Esomeprazole Magnesium — PPI compared to H2RA
  Other Names: Ranitidine

SUMMARY:
The principal investigator hypothesizes that participants receiving NSAID drugs with dyspeptic symptoms have increased production of gastric levels of free radicals. The primary objective of the study is to determine if Esomeprazole Magnesium increases gastric total antioxidant capacity and decreases gastric free radical production in humans. Participants (age 18 years and older) with no history of upper GI bleeding who are receiving non-steroidal anti-inflammatory drugs and then develop dyspepsia will be recruited from our primary care clinic in Washington, DC. All eligible participants will undergo biopsies of antrum and corpus. The participants will be randomized to receive either Zantac OTC or Nexium for 15 days. On day 15, all participants will undergo repeat upper endoscopy to obtain biopsies of antrum and corpus. Tissue samples will then be extracted to determine total antioxidant capacity and lipid peroxide levels (as an indirect marker of free radical production).

DETAILED DESCRIPTION:
An extensive meta-analysis has confirmed that dyspeptic symptoms are common in individuals using non-steroidal anti-inflammatory drugs (NSAIDs) (1). Both esomeprazole 20 mg daily and esomeprazole 40 mg daily have been shown to be more effective than placebo for the control of upper gastrointestinal symptoms in patients receiving NSAIDs (2).

The mechanisms by which H, K-ATPase inhibitors protect against NSAID gastropathy remain unclear, although it is known that their use is more clinically effective than the use of the H2-receptor antagonist, ranitidine (3).

The biochemical basis for NSAID gastropathy is not fully understood (6). One potential mechanism for the development of gastric damage in individuals receiving NSAIDs is oxidative stress related to depletion of gastric antioxidants. A recent endoscopic study in patients supports the hypothesis that NSAID use associated with gastric bleeding decreases gastric mucosal glutathione levels (7), a major cellular micronutrient antioxidant produced by mammalian cells. The principal investigator has been working on the possibility that activation of afferent nerve fibers by oxidative stress can induce abdominal discomfort during the use of NSAIDs. This notion is supported by animal studies that have shown that oxidants evoke neurotransmitter release from enteric neurons (8). This experimental result suggests that abnormal tissue levels of oxygen-derived free radicals (oxidative stress) could directly activate afferent enteric nerves or could alter gastric motility via a neuronal mechanism.

The hypothesis of this present proposal is that participants receiving NSAID drugs with dyspeptic symptoms have increased production of gastric levels of free radicals. The primary aims of this study are to examine gastric free radical production and total antioxidant capacity in participants who are taking NSAID drugs and have dyspeptic symptoms. Gastric free radical production and total antioxidant capacity will be measured before and after receiving either 15 days of daily esomeprazole magnesium or ranitidine.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are capable of providing informed consent, ages 18 years old and older. Partipants who are taking non-steroidal anti-inflammatory drugs on a daily basis must present with at least a 1 week history of dyspeptic symptoms including epigastric or upper abdominal discomfort or pain.

Exclusion Criteria:

* Participants presenting with only a complaint of heartburn will be excluded. Participants with alarm symptoms of vomiting, evidence of bleeding, inadvertent weight loss, or dysphagia will be excluded. Participants will be excluded if they have had upper endoscopy within 6 months prior to randomization. At the initial visit, participants will have a Helicobacter pylori IgG serology drawn and all participants with a positive serology will be excluded. Participants with a previous history of myocardial infarction, cerebrovascular infarction, gastric or duodenal ulcer disease, or carcinoma will be excluded. The study will not enroll participants who have received a H, K-ATPase inhibitor within the past 2 weeks. At the initial upper endoscopy, all participants with esophageal ulcer, esophageal cancer, gastric ulcer, gastric cancer, and duodenal ulcer will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12 (Estimated); Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
gastric levels of total antioxidant capacity and gastric lipid peroxide levels on Day 22 | 1 week
  Measurement of tissue levels in stomach biopsies of total antioxidant capacity (in nmole of Trolox equivalent/g wet tissue) and lipid peroxides (in nmole/g wet tissue).

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Koch, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Ofman JJ, Maclean CH, Straus WL, Morton SC, Berger ML, Roth EA, Shekelle PG. Meta-analysis of dyspepsia and nonsteroidal antiinflammatory drugs. Arthritis Rheum. 2003 Aug 15;49(4):508-18. doi: 10.1002/art.11192. PMID 12910557
- [Background] Hawkey C, Talley NJ, Yeomans ND, Jones R, Sung JJ, Langstrom G, Naesdal J, Scheiman JM; NASA1 SPACE1 Study Group. Improvements with esomeprazole in patients with upper gastrointestinal symptoms taking non-steroidal antiinflammatory drugs, including selective COX-2 inhibitors. Am J Gastroenterol. 2005 May;100(5):1028-36. doi: 10.1111/j.1572-0241.2005.41465.x. PMID 15842575
- [Background] Yeomans ND, Tulassay Z, Juhasz L, Racz I, Howard JM, van Rensburg CJ, Swannell AJ, Hawkey CJ. A comparison of omeprazole with ranitidine for ulcers associated with nonsteroidal antiinflammatory drugs. Acid Suppression Trial: Ranitidine versus Omeprazole for NSAID-associated Ulcer Treatment (ASTRONAUT) Study Group. N Engl J Med. 1998 Mar 12;338(11):719-26. doi: 10.1056/NEJM199803123381104. PMID 9494148
- [Background] Koch TR, Petro A, Darrabie M, Opara EC. Effect of the H, K-ATPase inhibitor, esomeprazole magnesium, on gut total antioxidant capacity in mice. J Nutr Biochem. 2004 Sep;15(9):522-6. doi: 10.1016/j.jnutbio.2004.03.003. PMID 15350983
- [Background] Koch TR, Petro A, Darrabie M, Opara EC. Effects of esomeprazole magnesium on nonsteroidal anti-inflammatory drug gastropathy. Dig Dis Sci. 2005 Jan;50(1):86-93. doi: 10.1007/s10620-005-1283-z. PMID 15712643
- See also: Related Info — http://www.medstarresearch.org